CLINICAL TRIAL: NCT04203238
Title: Meat and Potato Diet for Enhancing Cardiometabolic Health in Adults
Brief Title: Potato Research for Enhancing Metabolic Outcomes
Acronym: PREMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Principal Investigator, John Kirwan, Executive Director, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PBRC 2019-029
Record Dates: First submitted 2019-08-16; First posted 2019-12-18 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Insulin Resistance; Obesity
MeSH Terms: conditions — Insulin Resistance; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized parallel design
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator and care providers will be blinded to randomization and treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potatoes Lean Meat (PLM) (Experimental): The main entrée in the PLM arm will consist of a menu item in which 40% of the meat in the original recipe will be replaced with potatoes. The diet is designed to provide six or less ounces of meat/day which is consistent with the DASH diet.
  Interventions: Other: Reduced Meat High Potato Diet
- Lean Meat Pulses (LMP) (Experimental): The main entrée in the LMP arm will consist of a menu item in which 40% of the meat in the original recipe will be replaced with pulses. The diet is designed to provide six or less ounces of meat/day which is consistent with the DASH diet.
  Interventions: Other: Reduced Meat High Pulses Diet

INTERVENTIONS:
Other: Reduced Meat High Potato Diet — The main entrée in the PLM arm will consist of a menu item in which 40% of the meat in the original recipe will be replaced with potatoes.
  Arms: Potatoes Lean Meat (PLM)
Other: Reduced Meat High Pulses Diet — The main entrée in the LMP arm will consist of a menu item in which 40% of the meat in the original recipe will be replaced with pulses.
  Arms: Lean Meat Pulses (LMP)

SUMMARY:
The potato is a nutritious food that comprises approximately 30% of total vegetable intake in the United States (US). Consumption of pulses in the US is low but its contribution to health is frequently promoted. However, in the US diet, potatoes contribute as much dietary fiber, far more potassium, and a host of similar nutrients as pulses. When prepared to enhance its slowly digested starch content, potatoes produce a moderate glycemic response. In encouraging a shift towards plant-based foods and sustainable diets, the potato can partially replace meat in meat dishes to enhance the overall quality of the diet and reduce meat intake to recommended levels.

DETAILED DESCRIPTION:
Approximately 11% of individuals with untreated prediabetes progress to diabetes every year. Reversion to normal blood glucose concentrations reduces the incidence of diabetes by 56%. Healthy eating patterns such as the DASH and the Mediterranean Diet have shown that high intakes of fruits, vegetables, whole grains, legumes or pulses, and potatoes are associated with cardiometabolic health. In contrast, dietary patterns rich in meat and sugar-rich foods are associated with increased risk of mortality, type 2 diabetes, and coronary heart disease. These findings suggest that it may be prudent to replace certain foods with fruits and vegetables rather than simply embrace plant-based diets. Small changes that bestow health benefits are likely to be sustainable in the long-term. The objective of the present application is to develop a diet intervention to reverse insulin resistance in an overweight or obese population. The central hypothesis is that in the context of an overall healthy eating pattern, potatoes and pulses will not differ in the glycemic and insulinemic responses, lipid profile, and hsCRP concentration they elicit.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 - 60 years of age
* Body mass index between 25 and 40 kg/m2
* No evidence of diabetes (fasting blood sugar <126 mg/dL).
* HOMA-IR > 2
* Willing to consume the study foods and refrain from eating other foods for eight weeks.

Exclusion Criteria:

* Have type 1 or type 2 diabetes currently being treated by medication.
* Are being treated with medications that have a significant effect on insulin resistance, obesity, serum lipids, and metabolic rate, or medications that significantly increase body weight such as certain antidepressants, second-generation antipsychotics, systemic glucocorticoids, and adrenergic blockers or stimulators.
* Current pregnancy or breastfeeding.
* Women of childbearing potential who are not using an effective method of birth control (i.e., barrier method, intrauterine and cervical devices, oral contraceptives, hormonal injections (Depo Provera® ), condoms with spermicidal gel or foam, contraceptive patch (Ortho Evra), diaphragm, or abstinence), are not surgically sterilized (including tubal ligation and hysterectomy), or not at least two years postmenopausal. All women of childbearing potential will have a pregnancy test performed prior to starting the study treatment in each cohort. If a subject becomes pregnant during the study, they will be dropped from the study.
* Have clinically significant abnormal laboratory markers (as determined by the medical investigator).
* Have contraindications to participation in a diet intervention.
* Are unable to provide a baseline blood sample.
* Have any condition that impedes testing of the study hypothesis or makes it unsafe to consume the foods being tested in the study (determined by the investigative team).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kirwan, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rebello CJ, Beyl RA, Greenway FL, Atteberry KC, Hoddy KK, Kirwan JP. Low-Energy Dense Potato- and Bean-Based Diets Reduce Body Weight and Insulin Resistance: A Randomized, Feeding, Equivalence Trial. J Med Food. 2022 Dec;25(12):1155-1163. doi: 10.1089/jmf.2022.0072. Epub 2022 Nov 11. PMID 36367708

RESULTS

PARTICIPANT FLOW:
Groups:
- Lean Meat Pulses (LMP): The main entrée in the LMP arm will consist of a menu item in which 40% of the meat in the original recipe will be replaced with pulses. The diet is designed to provide six or less ounces of meat/day.
  Reduced Meat High Pulses Diet: The main entrée in the LMP arm will consist of a menu item in which 40% of the meat in the original recipe will be replaced with pulses.
Period: Overall Study
Arm/Group | Potatoes Lean Meat (PLM) | Lean Meat Pulses (LMP)
Started | 18 | 18
Completed | 14 | 17
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Covid-19 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Potatoes Lean Meat (PLM) | Lean Meat Pulses (LMP) | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years and standard error] | 44.6 (2.6) | 45.4 (2.6) | 45 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 12 | 23
  Non-White | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Response to the Diet
Description: Change in area under the curve for blood glucose (mg/dL/min) concentration in response to the diet. Negative values are considered a better outcome.
Time Frame: Baseline and 8 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL/min
Arm/Group | Potatoes Lean Meat (PLM) | Lean Meat Pulses (LMP)
Number analyzed (Participants) | 18 | 18
mg/dL/min | -103.44 (430.04) | -501.91 (406.83)

2. Secondary Outcome: Insulin Response to the Diet
Description: change in area under the curve for blood insulin (uU/mL/min) concentration in response to the diet. Negative values are considered a better outcome.
Time Frame: Baseline and 8 weeks
Measure: Least Squares Mean (Standard Error); unit: uU/ml/min
Groups:
- Potatoes Lean Meat (PLM): The main entrée in the PLM arm will consist of a menu item in which 40% of the meat in the original recipe will be replaced with potatoes. The diet is designed to provide six or less ounces of meat/day.
  Reduced Meat High Potato Diet: The main entrée in the PLM arm will consist of a menu item in which 40% of the meat in the original recipe will be replaced with potatoes.
Arm/Group | Potatoes Lean Meat (PLM) | Lean Meat Pulses (LMP)
Number analyzed (Participants) | 18 | 18
uU/ml/min | -966.63 (1012.49) | -2136.32 (955.53)

3. Secondary Outcome: Cholesterol Response to the Diet
Description: change in blood cholesterol (mg/dL) concentration in response to the diet. Negative values are considered a better outcome.
Time Frame: Baseline and 8 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Potatoes Lean Meat (PLM) | Lean Meat Pulses (LMP)
Number analyzed (Participants) | 18 | 18
mg/dL | -5.01 (3.57) | -11.79 (3.25)

4. Secondary Outcome: Triglyceride Response to the Diet
Description: change in blood triglyceride (mg/dL) concentration in response to the diet. Negative values are considered a better outcome.
Time Frame: Baseline and 8 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Potatoes Lean Meat (PLM) | Lean Meat Pulses (LMP)
Number analyzed (Participants) | 18 | 18
mg/dL | -4.67 (19.25) | -2.88 (17.94)

5. Secondary Outcome: LDL Particle Size Response to the Diet
Description: change in LDL particle size (nm) in response to the diet. Negative values are considered a better outcome.
Time Frame: Baseline and 8 weeks
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Potatoes Lean Meat (PLM) | Lean Meat Pulses (LMP)
Number analyzed (Participants) | 18 | 18
nm | -0.27 (0.13) | -0.38 (0.12)

6. Secondary Outcome: hsCRP Response to the Diet
Description: change in hsCRP (mg/L) in response to the diet. Positive values are considered a worse outcome.
Time Frame: Baseline and 8 weeks
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Potatoes Lean Meat (PLM) | Lean Meat Pulses (LMP)
Number analyzed (Participants) | 18 | 18
mg/L | 0.51 (1.43) | 0.24 (1.32)
Statistical Analysis 1: Comparison: Potatoes Lean Meat (PLM) vs Lean Meat Pulses (LMP); Test type: Superiority; p < 0.05, Mixed Models Analysis; Median Difference (Final Values) = 0.89

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Potatoes Lean Meat (PLM) | Lean Meat Pulses (LMP)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Potatoes Lean Meat (PLM) (N=18) | Lean Meat Pulses (LMP) (N=18)
gastrointestinal (Gastrointestinal disorders) | 0 (0) | 2 (2) — Two participants in the Bean diet group reported mild to moderate gastrointestinal effects (flatulence, cramps, and diarrhea). These effects resolved and participants completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT04203238/Prot_SAP_000.pdf